CLINICAL TRIAL: NCT00367458
Title: A Randomized Placebo Controlled Trial of Atorvastatin in HIV Positive Patients Not on Antiretroviral Medications With the Specific Aims of Studying the Effects of Atorvastatin on HIV Viral Load and Immune Activation Markers
Brief Title: Randomized Placebo-Controlled Trial of Atorvastatin in HIV-Positive Patients Not on Antiretroviral Therapy
Acronym: STATIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Frank Maldarelli, M.D., Staff Physician, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 060197; 06-I-0197 (Other: NIAID IRB); NCT00923546 (obsolete NCT alias)
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: HIV
Keywords: Viremia; Statin; HIV Replication; Cholesterol; Lipid Raft; HIV Infection; HIV Positive
MeSH Terms: conditions — Viremia; HIV Infections; HIV Seropositivity | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atorvastatin, then Placebo (Experimental): Patients were randomized to receive Atorvastatin first for 8 weeks, followed by 4 weeks wash out, and then cross over to placebo for 8 weeks.
  Interventions: Drug: Atorvastatin; Drug: Placebo
- Placebo, Then Atorvastatin (Experimental): Patients were randomized to receive placebo first for 8 weeks, followed by 4 weeks wash out, and then cross over to 80 mg atorvastatin daily for 8 weeks.
  Interventions: Drug: Atorvastatin; Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 80 mg atorvastatin oral daily
  Other Names: lipitor
Drug: Placebo — patients will be administered placebo
  Other Names: no other name for placebo

SUMMARY:
This study will examine the effects of atorvastatin, a statin (drug that lowers cholesterol) on the human immunodeficiency virus (HIV). If not treated, HIV infection causes an incurable, progressive deficiency in the immune system that leads to death, usually from disease that takes advantage of weakened immunity. Previous studies, however, have suggested that if the amount of cholesterol in infected cells is reduced, multiplication of HIV is also reduced. In this study, researchers will examine the HIV viral loads, that is, amount of the virus in the blood. They will evaluate the composition of the strain of the virus that patients carry (HIV genotype), response of the immune system to the virus, and how genes may determine the way in which the drug may or may not work against the strain of virus. Researchers plan to enroll 22 participants, anticipating a study to last 30 weeks for each participant.

Patients ages 18 or older with HIV infection, who are not pregnant or breastfeeding, who do not have a known allergy to atorvastatin use, and who have not had a serious illness or infection that required hospitalization within the 30 days before entering the study may be eligible for this study. They will be assigned to random groups: one that to receive atorvastatin and the other to receive a placebo, which has no effect on cholesterol or ability of the HIV infection to multiply. Patients will remain in their groups and treatments for 8 weeks. At the completion of 8 weeks, no matter the study group, all patients will be required to discontinue all study-related medications for 4 weeks. After that period, the study assignments will be switched, so that those previously taking the placebo will take atorvastatin, and vice versa. The study will proceed for another 8 weeks, followed by a period of stopping study-related medications and patients being observed for 4 weeks. Throughout the study, patients will have regularly scheduled visits at the clinic. At those visits there will be collection of blood samples, assessments of symptoms, physical examinations, and questionnaires to complete. Blood tests may require fasting beforehand, and blood samples will be used in standard tests, including those regarding the liver, kidneys, muscles, blood cells, and pregnancy status. Specialized blood tests will determine viral load, effects of the drug on the immune cells, and genetic influence on the drug's effectiveness.

DETAILED DESCRIPTION:
This protocol is a randomized, double blind, placebo controlled trial designed to study the effects of the lipid lowering statin, atorvastatin on HIV-1 viremia.

Untreated HIV-1 infection results in an incurable, progressive immunodeficiency and death, usually from opportunistic infections. Combination antiretroviral therapy (ARV) has been successful in suppressing HIV replication and reducing morbidity and mortality. Long term ARV therapy is associated with the development of HIV-1 drug resistance, and significant adverse side effects including metabolic and cardiovascular complications. Prolonged therapy with certain antiretrovirals is associated with increased risk of cardiovascular disease and a number of dyslipidemic syndromes, including increased levels of cholesterol, LDL, and triglycerides in peripheral blood. New therapeutic strategies to suppress HIV-1 infection are essential.

Previously, in vitro studies suggested that exposure to cholesterol-lowering statins results in decreases in HIV-1 replication. The mechanisms of inhibition remain uncertain, but possibilities include disrupting membrane trafficking or cytoskeletal processes necessary for intracellular transport of viral proteins, or altering cellular activation state necessary for viral gene expression. Initial in vivo studies of the effects of statins on HIV-1 have been largely anecdotal in nature and have yielded conflicting results. Although statin therapy is commonly used in HIV-1 infection, adverse effects from the combination of antiretrovirals and statins are possible. A more thorough understanding of the effects of statins on HIV-1 replication is essential to determine the potential therapeutic effect and to investigate the risks and benefits of this approach in vivo.

We plan to conduct a double blind randomized placebo controlled trial, with a cross over design, to study the effects of atorvastatin in 22 HIV-infected patients not currently taking antiretroviral therapy. Patients will be randomized to receive either placebo or atorvastatin 80mg for 8 weeks. After a 4-week wash out period patients on the atorvastatin arm will crossover to placebo and, vice versa patients in the placebo arm will cross over to atorvastatin for an additional 8 weeks. Upon completion of study medications all patients will be followed for 4 weeks. Each arm will have a minimum of 11 patients each. The primary outcome measure in this study is the effect of lipid lowering agents on HIV-1 RNA levels; additional secondary outcome measures include effects of lipid lowering agents on lipid profile, markers of inflammation and immune activation and investigations of host and viral genetic factors.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adults 18 years of age or older.
* Human Immunodeficiency Virus -1 (HIV-1) infection, as documented by a licensed Enzyme-Linked Immunosorbent Assay (ELISA) test kit and confirmed by a Western blot assay at any time point prior to study entry or at study entry (May do after informed consent if no test results are available).

Off all antiretroviral (ARV) for greater than or equal to three months prior to study entry, no documented evidence of viral resistance, and no evidence of acute HIV infection.

* Willingness to use a method of contraception during the study period.
* Willingness to have blood drawn.
* No known allergy or contraindication to atorvastatin use.
* Ability to understand and willingness to sign the informed consent.
* Willingness to have blood stored for future phenotyping and genotyping.
* Cluster of differentiation 4 (CD4) cell count greater than 350 cells/ml.
* 3 viral loads that average greater than 1000 copies/ml within a 4-week period.
* The viral loads will be done using the branched deoxyribonucleic acid (bDNA) method in the National Institutes of Health (NIH) laboratory and must be within 20% (log10bDNA of each other).
* A fasting total cholesterol lower than 240mg/dl and an Low-density lipoprotein (LDL) cholesterol lower than 130mg/dl.
* Liver function tests (aspartate aminotransferase (AST) or alanine aminotransferase (ALT)) not greater than 1.5 times the upper limit of normal.
* Creatine phosphokinase elevations (CPK) not greater than 3 times the upper limit of normal (ULN) on two sequential determinations and, in the opinion of the investigator, without clear association with exercise.
* Laboratory values:

Absolute neutrophil count (ANC) greater than or equal to 1000/mm(3).

Hemoglobin greater than or equal to 11.0 g/dL.

Platelet count greater than or equal to 100,000/mm(3).

Creatinine less than or equal to 2 x ULN.

Serum amylase and lipase less than or equal to 1.25 x ULN.

* Negative serum pregnancy test at randomization.

EXCLUSION CRITERIA:

* Pregnancy or breast feeding.
* Active drug use or alcohol abuse/dependence, which in the opinion of the investigators, will interfere with the patient's ability to participate in the study.
* Serious illness requiring systemic treatment and/or hospitalization within 30 days of entry.
* Evidence of active opportunistic infections or neoplasms that require chemotherapy during the study period except cutaneous Kaposi Sarcoma.
* Allergy or hypersensitivity to atorvastatin or any of its components.
* History of myositis or rhabdomyolysis with use of any statins.
* History of inflammatory muscle disease such as poly or dermatomyositis.
* Concomitant use of fibric acid derivatives or other lipid lowering agents including patients on statins and Ezetimibe.
* Concomitant use of drugs that have significant interactions with atorvastatin. Please see appendix II for a listing.
* Concomitant use of St.Johns wort.
* Concomitant use of Valproic acid.
* Patients who are on concurrent immunomodulatory agents, including systemic corticosteroids, will be ineligible for 3 months after completion of therapy with the immunomodulating agents. Topical, nasal or inhaled corticosteroids use is not an exclusion criterion.
* Serum LDL cholesterol less than 40 mg/dl.
* Vaccinations within 6 weeks of study entry.
* Vaccinations within 6 weeks of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-10-18 (Actual); Primary Completion 2008-06-19 (Actual); Study Completion 2008-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Maldarelli, M.D. Ph.D., Principal Investigator — National Cancer Institute (NCI), National Institutes of Health (NIH)
Locations (3):
- United States (3):
  - Naval Medical Center, San Diego, San Diego, California
  - National Naval Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palella FJ Jr, Delaney KM, Moorman AC, Loveless MO, Fuhrer J, Satten GA, Aschman DJ, Holmberg SD. Declining morbidity and mortality among patients with advanced human immunodeficiency virus infection. HIV Outpatient Study Investigators. N Engl J Med. 1998 Mar 26;338(13):853-60. doi: 10.1056/NEJM199803263381301. PMID 9516219
- [Background] Carr A, Cooper DA. Adverse effects of antiretroviral therapy. Lancet. 2000 Oct 21;356(9239):1423-30. doi: 10.1016/S0140-6736(00)02854-3. PMID 11052597
- [Background] Carr A, Samaras K, Thorisdottir A, Kaufmann GR, Chisholm DJ, Cooper DA. Diagnosis, prediction, and natural course of HIV-1 protease-inhibitor-associated lipodystrophy, hyperlipidaemia, and diabetes mellitus: a cohort study. Lancet. 1999 Jun 19;353(9170):2093-9. doi: 10.1016/S0140-6736(98)08468-2. PMID 10382692

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin First, Then Placebo: Patients were randomized to receive Atorvastatin first for 8 weeks, followed by 4 weeks wash out, and then cross over to placebo for 8 weeks.
- Placebo First, Then Atorvastatin: Patients were randomized to receive placebo first for 8 weeks, followed by 4 weeks wash out, and then cross over to 80 mg atorvastatin daily for 8 weeks.
Period: First Intervention - 8 Weeks
Arm/Group | Atorvastatin First, Then Placebo | Placebo First, Then Atorvastatin
Started | 12 | 12
Completed | 10 | 12
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0
Period: Washout Period - 4-6 Weeks
Arm/Group | Atorvastatin First, Then Placebo | Placebo First, Then Atorvastatin
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0
Period: Second Intervention - 8 Weeks
Arm/Group | Atorvastatin First, Then Placebo | Placebo First, Then Atorvastatin
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin First, Then Placebo | Placebo First, Then Atorvastatin | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 30 [21 to 46] | 30 [21 to 46] | 30 [21 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Human Immunodeficiency Virus 1 (HIV-1) Ribonucleic Acid (RNA) Levels
Description: The change in HIV viral RNA level in plasma in response to lipid lowering agents was measured as log10 plasma RNA copy number, and the change in the log10 viral RNA level is included in table.
Time Frame: Baseline and 8 weeks
Measure: Median (Inter-Quartile Range); unit: Log10 copies/ml plasma
Groups:
- Atorvastatin: Patients were randomized to receive Atorvastatin for 8 weeks
- Placebo: Patients were randomized to receive placebo for 8 weeks
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 24 | 24
Log10 copies/ml plasma
  Baseline | 0 [0 to 0] | 0 [0 to 0]
  8 Weeks | -0.03 [-0.35 to 0.04] | -0.08 [-0.25 to 0.08]

2. Secondary Outcome: Change in Percentage of Cluster of Differentiation 4 (CD4+) Human Leukocyte Antigen DR (HLA-DR+) in Peripheral Blood
Description: CD4+HLA-DR+ are cellular markers of immune activation that is present in HIV infected individuals. This marker was measured before and after the statin/placebo intervention by standard lymphocyte phenotyping.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: percent T cell subset
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 24 | 24
percent T cell subset
  Baseline CD4+HLA-DR+ | 0 (5.34) | 0 (7.35)
  CD4+HLA-DR+ at 8 Weeks | -2 (5.05) | -1.8 (10.2)

3. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 26 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 24 | 24
Participants | 12 | 12

4. Secondary Outcome: Change in Percentage of Cluster of Differentiation 8 (CD8+) Human Leukocyte Antigen DR (HLA-DR+) in Peripheral Blood
Description: CD8+HLA-DR+ are cellular markers of immune activation that is present in HIV infected individuals. This marker was measured before and after the statin/placebo intervention by standard lymphocyte phenotyping.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: percent T cell subset
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 24 | 24
percent T cell subset
  Baseline CD8+HLA-DR+ | 0 (10.28) | 0 (12.52)
  CD8+HLA-DR+ at 8 Weeks | -3.8 (8.80) | -3.5 (12.15)

5. Secondary Outcome: Change in Percentage of Cluster of Differentiation 8 (CD8+) Human Leukocyte Antigen DR (HLA-DR+), CD8+(CD8+HLADR+CD38+) in Peripheral Blood
Description: CD8+HLADR+CD38+ are cellular markers of immune activation that is present in HIV infected individuals. This marker was measured before and after the statin/placebo intervention by standard lymphocyte phenotyping.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: percent T cell subset
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 24 | 24
percent T cell subset
  Baseline CD8+HLADR+CD38+ | 0 (12.31) | 0 (11.01)
  CD8+HLADR+CD38+ at 8 Weeks | -3.75 (10.37) | -3.3 (13.28)

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 26 weeks
Arm/Group | Atorvastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/24 | 2/24
Other Adverse Events (participants affected / at risk) | 12/24 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=24) | Placebo (N=24)
low LDL (Metabolism and nutrition disorders) | 2 (2) | 2 (2) — Due to concerns about the safety of intense lipid lowering in animal models, we established pre-specified LDL-c level (i.e., LDL-c<40 mg/dl) for early termination
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=24) | Placebo (N=24)
Abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Cardiac disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Herpes simplex (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flush (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Supplementation therapy (Surgical and medical procedures) | 1 (1) | 0 (0) — Dietary supplement
Treponema test positive (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2007-09-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT00367458/Prot_SAP_000.pdf
  • Informed Consent Form: Standard consent (2008-03-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT00367458/ICF_001.pdf
  • Informed Consent Form: Screening consent (2008-03-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT00367458/ICF_002.pdf